CLINICAL TRIAL: NCT05186805
Title: Open Label Maximal Use Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Tapinarof Cream, 1% in Pediatric Subjects With Extensive Atopic Dermatitis
Brief Title: Maximal Use Study of Tapinarof Cream, 1% in Pediatric Subjects With Extensive Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMVT-505-2104
Record Dates: First submitted 2021-11-08; First posted 2022-01-11 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis
Keywords: eczema; pediatric; tapinarof; phase 2; topical
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- tapinarof cream (Experimental): Tapinarof (DMVT-505) cream, 1% applied topically once daily
  Interventions: Drug: Tapinarof cream, 1%

INTERVENTIONS:
Drug: Tapinarof cream, 1% — Tapinarof cream, 1% applied topically once daily
  Other Names: DMVT-505

SUMMARY:
This is an open-label, multicenter study to evaluate the systemic exposure and safety of topical tapinarof cream, 1% under conditions of maximal use in pediatric subjects with atopic dermatitis

DETAILED DESCRIPTION:
This is a 4-week open-label study in which subjects will be assigned to receive tapinarof cream, 1% once daily for 4 weeks. At the end of the 4-week study treatment, qualified subjects will have the option to enroll in an open-label, long-term extension study for an additional 48 weeks of treatment. Subjects who do not participate in the open-label, long-term extension study will complete a follow-up visit approximately one week after the end of treatment in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects age 2 to 17 with a confirmed clinical diagnosis of atopic dermatitis and present for at least 6 months for ages 6-17 years old, 3 months for ages 2-5 years old
* BSA involvement ≥ 25% for subjects ages 12-17 years old, or ≥ 35% for subjects ages 2-11 years old, suitable for topical therapy.
* vIGA-AD score of ≥ 3 at screening and baseline (pre-dose)
* Female subjects of child bearing potential who are engaging in sexual activity that could lead to pregnancy agree to follow the specified contraceptive guidance throughout the study
* Capable of giving written informed consent
* Negative pregnancy test at Baseline (Day 1)

Exclusion Criteria:

* Immunocompromised at screening
* Chronic or acute systemic or superficial infection requiring treatment with systemic antibacterials or antifungals within one week prior to baseline visit
* Significant dermatological or inflammatory condition other than AD that, in the Investigator's opinion, would make it difficult to interpret data or assessments during the study
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥2.0x the upper limit of normal (ULN).
* Screening total bilirubin > 1.5x ULN
* Current or chronic history of liver disease
* Current or history of cancer within 5 years except for adequately treated cutaneous basal cell carcinoma, squamous cell carcinoma or carcinoma in situ of the cervix
* Subjects who would not be considered suitable for topical therapy
* Use of any prohibited medication or procedure within the indicated period before the baseline visit including other investigational product within 30 days or 5 half-lives of the investigational product (whichever is longer)
* History of or ongoing serious illness or medical, physical, or psychiatric condition(s) that, in the Investigator's opinion, may interfere with the subject's participation in the study, interpretation of results, or ability to understand and give informed consent.
* Pregnant or lactating females
* History of sensitivity to the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the -Investigator or Medical Monitor, contraindicates their participation
* Previous known participation in a clinical study with tapinarof (previously known as GSK2894512 and WBI-1001)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Villalobos, Study Director — Dermavant Sciences, Inc.
Locations (10):
- United States (9):
  - Dermavant Investigative Site, Thousand Oaks, California
  - Dermavant Investigative Site, Centennial, Colorado
  - Dermavant Investigative Site, Coral Gables, Florida
  - Dermavant Investigative Site, Hialeah, Florida
  - Dermavant Investigative Site, Miami Lakes, Florida
  - Dermavant Investigative Site, Chicago, Illinois
  - Dermavant Investigative Site, Summerville, South Carolina
  - Dermavant Investigative Site, Houston, Texas
  - Dermavant Investigative Site, San Antonio, Texas
- Dermavant Investigative Site, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bashaw ED, Tran DC, Shukla CG, Liu X. Maximal Usage Trial: An Overview of the Design of Systemic Bioavailability Trial for Topical Dermatological Products. Ther Innov Regul Sci. 2015 Jan;49(1):108-115. doi: 10.1177/2168479014539157. Epub 2014 Jun 27. PMID 26634191
- [Background] Bieber T. Atopic dermatitis. N Engl J Med. 2008 Apr 3;358(14):1483-94. doi: 10.1056/NEJMra074081. No abstract available. PMID 18385500
- [Background] Cappon GD and Hurtt ME. Developmental toxicity of the kidney. In: Kapp RW and Yyl L, editors. Reproductive Toxicology, Target Organ Series, 3rd edition. New York:Informa Healthcare, 2010:193-204.
- [Background] Carroll CL, Balkrishnan R, Feldman SR, Fleischer AB Jr, Manuel JC. The burden of atopic dermatitis: impact on the patient, family, and society. Pediatr Dermatol. 2005 May-Jun;22(3):192-9. doi: 10.1111/j.1525-1470.2005.22303.x. PMID 15916563
- [Background] Frazier KS and Seely JC. Urinary system. In: Sahota PS, Popp JA, Hardisty JF and Gopinath C, editors. Toxicologic Pathology. Nonclinical Safety Assessment. CRC Press, 2013:421-84.
- [Background] Furue M, Hashimoto-Hachiya A, Tsuji G. Aryl Hydrocarbon Receptor in Atopic Dermatitis and Psoriasis. Int J Mol Sci. 2019 Oct 31;20(21):5424. doi: 10.3390/ijms20215424. PMID 31683543
- [Background] Hanifin JM, Rajka G. Diagnostic features of atopic dermatitis. Acta Dermato-Venereologica Supplementum. 1980;92:44-7.
- [Background] Hanifin JM, Thurston M, Omoto M, Cherill R, Tofte SJ, Graeber M. The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. EASI Evaluator Group. Exp Dermatol. 2001 Feb;10(1):11-8. doi: 10.1034/j.1600-0625.2001.100102.x. PMID 11168575
- [Background] Kalia YN, Nonato LB, Lund CH, Guy RH. Development of skin barrier function in premature infants. J Invest Dermatol. 1998 Aug;111(2):320-6. doi: 10.1046/j.1523-1747.1998.00289.x. PMID 9699737
- [Background] Lewis-Jones S. Quality of life and childhood atopic dermatitis: the misery of living with childhood eczema. Int J Clin Pract. 2006 Aug;60(8):984-92. doi: 10.1111/j.1742-1241.2006.01047.x. PMID 16893440
- [Background] Nikolovski J, Stamatas GN, Kollias N, Wiegand BC. Barrier function and water-holding and transport properties of infant stratum corneum are different from adult and continue to develop through the first year of life. J Invest Dermatol. 2008 Jul;128(7):1728-36. doi: 10.1038/sj.jid.5701239. Epub 2008 Jan 17. PMID 18200056
- [Background] Peppers J, Paller AS, Maeda-Chubachi T, Wu S, Robbins K, Gallagher K, Kraus JE. A phase 2, randomized dose-finding study of tapinarof (GSK2894512 cream) for the treatment of atopic dermatitis. J Am Acad Dermatol. 2019 Jan;80(1):89-98.e3. doi: 10.1016/j.jaad.2018.06.047. Epub 2018 Jul 3. PMID 30554600
- [Background] Smith SH, Jayawickreme C, Rickard DJ, Nicodeme E, Bui T, Simmons C, Coquery CM, Neil J, Pryor WM, Mayhew D, Rajpal DK, Creech K, Furst S, Lee J, Wu D, Rastinejad F, Willson TM, Viviani F, Morris DC, Moore JT, Cote-Sierra J. Tapinarof Is a Natural AhR Agonist that Resolves Skin Inflammation in Mice and Humans. J Invest Dermatol. 2017 Oct;137(10):2110-2119. doi: 10.1016/j.jid.2017.05.004. Epub 2017 Jun 6. PMID 28595996
- [Background] Zoetis T, Hurtt ME. Species comparison of anatomical and functional renal development. Birth Defects Res B Dev Reprod Toxicol. 2003 Apr;68(2):111-20. doi: 10.1002/bdrb.10013. No abstract available. PMID 12866702
- [Derived] Paller AS, Hebert AA, Gonzalez ME, Butners V, Fitzgerald N, Tabolt G, Rubenstein DS, Piscitelli SC. Maximal Usage Trial of Tapinarof Cream 1% Once Daily in Pediatric Patients Down to 2 Years of Age with Extensive Atopic Dermatitis. Am J Clin Dermatol. 2025 May;26(3):449-456. doi: 10.1007/s40257-025-00929-9. Epub 2025 Mar 24. PMID 40126804

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from the DMVT-505-2104 study had the option to participate in the open label extension study (DMVT-505-3103, NCT05142774).
Period: Overall Study
Arm/Group | Tapinarof Cream
Started | 36
Completed | 32
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.9 (4.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Validated Investigator Global Assessment for Atopic Dermatitis [Count of Participants; unit: Participants]
  0 - Clear | 0
  1 - Almost Clear | 0
  2 - Mild | 0
  3 - Moderate | 28
  4 - Severe | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experienced Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of Participants that Experienced Adverse Events (AEs) and Serious Adverse Events (SAEs).
Time Frame: Baseline to Day 28 for subjects enrolling in Long-Term Extension (LTE), otherwise to Day 35
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 36
Participants
  Experienced an AE | 8
  Experienced an SAE | 0

2. Primary Outcome: Change From Baseline in Laboratory Values (U/L)
Description: Change in laboratory values was assessed for clinical relevance
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 36
U/L
  Alanine aminotransferase (U/L): number analyzed (Participants) | 30
  Alanine aminotransferase (U/L) | 1.9 (10.80)
  Alkaline phosphatase (U/L): number analyzed (Participants) | 31
  Alkaline phosphatase (U/L) | 0.7 (52.95)
  Aspartate aminotransferase (U/L): number analyzed (Participants) | 30
  Aspartate aminotransferase (U/L) | 0.6 (6.44)

3. Primary Outcome: Change From Baseline in Laboratory Values (g/L)
Description: Change in laboratory values was assessed for clinical relevance
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 36
g/L
  Albumin (g/L): number analyzed (Participants) | 31
  Albumin (g/L) | -0.7 (2.72)
  Protein (g/L): number analyzed (Participants) | 31
  Protein (g/L) | -0.5 (4.20)
  Ery. mean corpuscular HGB Concentration (g/L): number analyzed (Participants) | 30
  Ery. mean corpuscular HGB Concentration (g/L) | -1.7 (7.68)
  Hemoglobin (g/L): number analyzed (Participants) | 30
  Hemoglobin (g/L) | 0.0 (7.61)

4. Primary Outcome: Change From Baseline in Laboratory Values (mmol/L)
Description: Change in laboratory values was assessed for clinical relevance
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 36
mmol/L
  Bicarbonate (mmol/L): number analyzed (Participants) | 31
  Bicarbonate (mmol/L) | -0.3 (2.16)
  Calcium (mmol/L): number analyzed (Participants) | 31
  Calcium (mmol/L) | -0.006 (0.0846)
  Chloride (mmol/L): number analyzed (Participants) | 31
  Chloride (mmol/L) | 0.0 (2.99)
  Glucose (mmol/L): number analyzed (Participants) | 29
  Glucose (mmol/L) | 0.20 (0.819)
  Potassium (mmol/L): number analyzed (Participants) | 29
  Potassium (mmol/L) | 0.08 (0.532)
  Sodium (mmol/L): number analyzed (Participants) | 31
  Sodium (mmol/L) | 0.1 (1.98)
  Blood urea nitrogen (mmol/L): number analyzed (Participants) | 31
  Blood urea nitrogen (mmol/L) | -0.06 (0.989)

5. Primary Outcome: Change From Baseline in Laboratory Values (Umol/L)
Description: Change in laboratory values was assessed for clinical relevance
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Mean (Standard Deviation); unit: Umol/L
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 36
Umol/L
  Bilirubin (umol/L): number analyzed (Participants) | 30
  Bilirubin (umol/L) | -0.34 (3.700)
  Enzymatic Creatinine (umol/L): number analyzed (Participants) | 30
  Enzymatic Creatinine (umol/L) | -0.9 (7.66)
  Urate (umol/L): number analyzed (Participants) | 31
  Urate (umol/L) | -6.0 (52.16)

6. Primary Outcome: Change From Baseline in Laboratory Values (10^9 Cells/L)
Description: Change in laboratory values was assessed for clinical relevance
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 36
10^9 cells/L
  Basophils (10^9/L): number analyzed (Participants) | 30
  Basophils (10^9/L) | 0.01 (0.048)
  Eosinophils (10^9/L): number analyzed (Participants) | 30
  Eosinophils (10^9/L) | 0.00 (0.419)
  Leukocytes (10^9/L) | 0.71 (2.451)
  Lymphocytes (10^9/L): number analyzed (Participants) | 30
  Lymphocytes (10^9/L) | 0.38 (1.095)
  Monocytes (10^9/L): number analyzed (Participants) | 30
  Monocytes (10^9/L) | -0.06 (0.175)
  Neutrophils (10^9/L): number analyzed (Participants) | 30
  Neutrophils (10^9/L) | 0.36 (2.124)
  Platelets (10^9/L): number analyzed (Participants) | 30
  Platelets (10^9/L) | -34.8 (95.27)

7. Primary Outcome: Change From Baseline in Laboratory Values (%)
Description: Change in laboratory values was assessed for clinical relevance
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Mean (Standard Deviation); unit: % of cells
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 36
% of cells
  Basophils/Total cells (%): number analyzed (Participants) | 30
  Basophils/Total cells (%) | 0.05 (0.343)
  Eosinophils/Total cells (%): number analyzed (Participants) | 30
  Eosinophils/Total cells (%) | -0.13 (4.606)
  Lymphocytes/Total cells (%): number analyzed (Participants) | 30
  Lymphocytes/Total cells (%) | 0.81 (11.023)
  Monocytes/Total cells (%): number analyzed (Participants) | 30
  Monocytes/Total cells (%) | -0.81 (2.662)
  Neutrophils/Total cells (%): number analyzed (Participants) | 30
  Neutrophils/Total cells (%) | 0.08 (12.693)
  Reticulocytes/Erythrocytes (%): number analyzed (Participants) | 29
  Reticulocytes/Erythrocytes (%) | 0.06 (0.377)

8. Primary Outcome: Change From Baseline in Laboratory Values (pg)
Description: Change in Ery. mean corpuscular hemoglobin laboratory values was assessed for clinical relevance
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 30
pg | 0.26 (0.787)

9. Primary Outcome: Change From Baseline in Laboratory Values (fL)
Description: Change in Ery. mean corpuscular volume laboratory values was assessed for clinical relevance
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 30
fL | 1.26 (1.973)

10. Primary Outcome: Change From Baseline in Laboratory Values (10^12 Cells/L)
Description: Change in Erythrocytes laboratory values was assessed for clinical relevance
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 30
10^12 cells/L | -0.055 (0.2481)

11. Primary Outcome: Change From Baseline in Laboratory Values (L/L)
Description: Change in Hematocrit laboratory values was assessed for clinical relevance
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Mean (Standard Deviation); unit: L/L
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 30
L/L | 0.002 (0.0228)

12. Primary Outcome: Mean Change in Local Tolerability Scale (LTS)
Description: Local Tolerability Scale (LTS) is a clinical tool for assessing the presence and overall degree of irritation at the application sites, according to a 5-point scale. 0 indicates no irritation and 4 indicates Very Severe irritation.
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 36
Units on a scale
  Baseline: number analyzed (Participants) | 35
  Baseline | 0.2 (0.68)
  Day 28: number analyzed (Participants) | 31
  Day 28 | 0.1 (0.40)

13. Primary Outcome: Tapinarof Plasma PK Parameters on Day 1: AUC0-τ
Description: The AUC in plasma is a pharmacokinetic parameter that describes the overall exposure of the drug.
Time Frame: Day 1 (PK samples collected pre-dose and at 1, 3, and 5 hours post-dose)
Population: PK population
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 34
pg*h/mL | 4690 (5600)

14. Primary Outcome: Tapinarof Plasma PK Parameters on Day 1: Cmax
Description: The Cmax is a pharmacokinetic parameter that describes the highest concentration of the drug that is achieved after dosing.
Time Frame: Day 1 (PK samples collected pre-dose and at 1, 3, and 5 hours post-dose)
Population: PK population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 35
pg/mL | 2440 (3900)

15. Primary Outcome: Tapinarof Plasma PK Parameters on Day 1: Tmax
Description: The tmax is a pharmacokinetic parameter that describes the time point at which the highest concentration of the drug is achieved after dosing.
Time Frame: Day 1 (PK samples collected pre-dose and at 1, 3, and 5 hours post-dose)
Population: PK population
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 34
hour | 2.37 (1.19)

16. Primary Outcome: Tapinarof Plasma Concentration: Cτ
Description: The Cτ is a pharmacokinetic parameter that is the last quantifiable concentration determined directly from individual concentration-time data
Time Frame: Day 1 (PK samples collected pre-dose and at 1, 3, and 5 hours post-dose)
Population: PK Population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 34
pg/mL | 1330 (3780)

17. Primary Outcome: Change From Baseline in Vital Signs (Beats/Min)
Description: Change in pulse vital signs was assessed for clinical relevance
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Mean (Standard Deviation); unit: Beats/Min
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 36
Beats/Min | 0.9 (14.40)

18. Primary Outcome: Change From Baseline in Vital Signs (mmHg)
Description: Change in Blood Pressure vital signs was assessed for clinical relevance
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 32
mmHg
  Systolic Blood Pressure (mmHg) | 1.1 (8.78)
  Diastolic Blood Pressure (mmHg) | -0.9 (6.63)

19. Primary Outcome: Change From Baseline in Vital Signs (C)
Description: Change in Temperature vital signs was assessed for clinical relevance
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Mean (Standard Deviation); unit: degrees C
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 32
degrees C | -0.08 (0.402)

20. Secondary Outcome: Change From Baseline in Validated Investigator Global Assessment in Atopic Dermatitis (vIGA-AD)
Description: The vIGA-AD is a global assessment of the current state of the disease. It is a static 5-point scale used to grade overall disease severity (scalp excluded), as determined by the investigator, using the clinical characteristics of erythema, induration/papulation, lichenification, oozing/crusting. The vIGA-AD ranges from 0 to 4 and is calculated as Clear (0), Almost clear (1), Mild (2), Moderate (3), and Severe (4). Higher vIGA-AD scores represent more severe disease.
Time Frame: Baseline to Day 28
Population: Safety population, Observed Cases
Measure: Count of Participants; unit: Participants
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 32
Participants
  +4 = worsened by 4 | 0
  +3 = worsened by 3 | 0
  +2 = worsened by 2 | 0
  +1 = worsened by 1 | 0
  0 - no change | 8
  -1 = improved by 1 | 14
  -2 = improved by 2 | 8
  -3 = improved by 3 | 2
  -4 = improved by 4 | 0

21. Secondary Outcome: Number of Subjects Who Have a Validated Investigator Global Assessment in Atopic Dermatitis (vIGA-AD) Score of Almost Clear (0 or 1) and at Least a 2-grade Reduction From Baseline
Description: as for outcome 20
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Count of Participants; unit: Participants
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 32
Participants | 8

22. Secondary Outcome: Number of Subjects With ≥50%, Improvement in Eczema Area and Severity Index (EASI) Score
Description: The Eczema Area and Severity Index (EASI) is a scoring system that takes into account the overall severity of disease based on lesion severity and the extent of percent body surface area affected with atopic dermatitis. The EASI is a composite score ranging from 0 -72 that takes into account the degree of erythema, edema/papulation, excoriation, and lichenification (each scored from 0 to 3 separately) for each of four body regions, with adjustment for the percent body surface area involved for each body region relative to the whole body. A higher EASI score represents more severe disease.
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Count of Participants; unit: Participants
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 32
Participants | 20

23. Secondary Outcome: Number of Subjects With ≥75%, Improvement in Eczema Area and Severity Index (EASI) Score
Description: The EASI is a composite score ranging from 0 to 72 that takes into account the degree of erythema, edema/papulation, excoriation, and lichenification (each scored from 0 to 3 separately) for each of four body regions, with adjustment for the %BSA involved for each body region relative to the whole body. Higher EASI scores indicate more severe disease.
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Count of Participants; unit: Participants
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 32
Participants | 7

24. Secondary Outcome: Number of Subjects With ≥90%, Improvement in Eczema Area and Severity Index (EASI) Score
Description: as for outcome 23
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Count of Participants; unit: Participants
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 32
Participants | 4

25. Secondary Outcome: Mean Change in Eczema Area and Severity Index EASI From Baseline to Day 28
Description: as for outcome 23
Time Frame: Baseline to Day 28
Population: Safety Population, Observed cases
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 32
scores on a scale | -12.16 (9.742)

26. Secondary Outcome: Percent Change in Eczema Area and Severity Index EASI From Baseline to Day 28
Description: as for outcome 23
Time Frame: Baseline to Day 28
Population: Safety Population, Observed cases
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 32
% change from baseline | -53.38 (38.337)

27. Secondary Outcome: Mean Change in Percent of Total Body Surface Area (%BSA) Affected
Description: The assessment of %BSA affected is an estimate of the percentage of total involved skin with psoriasis. For the purpose of clinical estimation, the total palmar surface of the subject's palm and digits may be assumed to be approximately equivalent to 1% BSA. The %BSA affected by psoriasis will be evaluated (from 0% to 100%). %BSA is a static assessment made without reference to previous scores.
Time Frame: Baseline to Day 28
Population: Safety Population, Observed cases
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 32
percentage of BSA | -21.06 (18.789)

28. Secondary Outcome: Percent Change in Percent of Total Body Surface Area (%BSA) Affected
Description: as for outcome 27
Time Frame: Baseline to Day 28
Population: Safety Population, Observed cases
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 32
% change from baseline | -49.40 (41.3000)

29. Secondary Outcome: Mean Change in Total Body Surface Area (BSA) x Validated Investigator Global Assessment in Atopic Dermatitis (vIGA-AD) Values
Description: The vIGA-AD is a clinical tool for assessing the current state/severity of a subject's atopic dermatitis at a given timepoint. It is a static 5-point morphological assessment of overall disease severity using the clinical characteristics of erythema, induration/papulation, lichenification, oozing/crusting (0 indicates no inflammatory signs of atopic dermatitis and 4 indicates disease is widespread). The assessment of %BSA affected is an estimate of the percentage of total involved skin with psoriasis. For clinical estimation, the total palmar surface of the subject's palm and digits may be assumed to be approximately equivalent to 1% BSA. %BSA is a static assessment made without reference to previous scores and will be evaluated 0-100%. The computation is referenced below, and no unit is applicable for this outcome measure. A negative change indicates improvement in disease.
  [Total Body Surface Area (BSA) x Validated Investigator Global Assessment in Atopic Dermatitis (vIGA-AD)]
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 32
unitless | -85.15 (65.848)

30. Secondary Outcome: Percent Change in Total Body Surface Area (BSA) x Validated Investigator Global Assessment in Atopic Dermatitis (vIGA-AD) Values
Description: The vIGA-AD is a clinical tool for assessing the current state/severity of a subject's atopic dermatitis at a given timepoint. It is a static 5-point morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema, induration/papulation, lichenification, oozing/crusting. Score of 0 indicates no inflammatory signs of atopic dermatitis and a 4 indicates disease is widespread in extent. The assessment of %BSA affected is an estimate of the percentage of total involved skin with psoriasis. For the purpose of clinical estimation, the total palmar surface of the subject's palm and digits may be assumed to be approximately equivalent to 1% BSA. The %BSA affected by psoriasis will be evaluated (from 0% to 100%). %BSA is a static assessment made without reference to previous scores.
  Computation: Total Body Surface Area (BSA) x Validated Investigator Global Assessment in Atopic Dermatitis (vIGA-AD)
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 32
% change from baseline | -62.77 (35.290)

31. Secondary Outcome: Mean Change in Average Weekly Peak Pruritus Numerical Rating Scale (PP-NRS) Score
Description: The PP-NRS is a scale from 0-10 used to assess itch/pruritus severity over a 24-hour period which will be used daily to assess peak pruritus. Higher PP-NRS ratings represent more itch reported.
Time Frame: Baseline to Day 28
Population: Safety Population, Observed Cases
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 33
Units on a scale | -4.155 (2.4558)

32. Secondary Outcome: Proportion of Subjects With a Baseline Peak Pruritus Numerical Rating Scale (PP-NRS) Score ≥4 Who Achieved ≥4-point Reduction in PP-NRS Score
Description: as for outcome 31
Time Frame: Baseline to Day 28
Population: Safety Population, Observed cases, subjects with baseline PP-NRS score ≥4
Measure: Count of Participants; unit: Participants
Arm/Group | Tapinarof Cream
Number analyzed (Participants) | 32
Participants
  Achieved ≥ 4-Point Reduction from Baseline in the Average Weekly PP-NRS Score | 14
  Failure to Achieve a ≥ 4-point Reduction from Baseline in the Average Weekly PP-NRS Score | 18

ADVERSE EVENTS:
Time Frame: Baseline to Day 28 for subjects enrolling in Long-Term Extension (LTE), otherwise to Day 35
Arm/Group | Tapinarof Cream
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 8/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tapinarof Cream (N=36)
Headache (Nervous system disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pustule (Infections and infestations) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Tranaminases increased (Investigations) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT05186805/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT05186805/SAP_001.pdf